CLINICAL TRIAL: NCT05660291
Title: Effects of Time Restricted Eating on Obesity: Comparing Windows of Eating to Achieve Weight Loss in Overweight and Obese Adults; a Pilot Study
Brief Title: A Study of Time Restricted Eating in Obese Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bradley A. Bohn, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-010547
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Overweight
Keywords: Body Mass Index (BMI) ≥ 25 kg/m^2; Early and late time-restricted eating
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early time-restricted eating (Experimental): Subjects window for eating would be between 08:00 AM - 4:00 PM
  Interventions: Behavioral: Early time-restricted eating
- Late time-restricted eating (Experimental): Subjects window for eating would be between 12:00 PM (noon) and 8:00 PM
  Interventions: Behavioral: Late time-restricted eating

INTERVENTIONS:
Behavioral: Early time-restricted eating — Subjects can eat whatever they want between the hours of 8:00 AM and 4:00 PM and can only consume water, black coffee/tea, or other zero calorie drinks (artificial sweeteners are okay) outside your designated eating window (from 4:00 PM to 8:00 AM).
  Arms: Early time-restricted eating
Behavioral: Late time-restricted eating — Subjects can eat whatever they want between the hours of 12:00 PM and 8:00 PM and can only consume water, black coffee/tea, or other zero calorie drinks (artificial sweeteners are okay) outside your designated eating window (from 8:00 PM to noon).
  Arms: Late time-restricted eating

SUMMARY:
The purpose of this pilot study is to understand the difference between early and late time-restricted eating on weight and body mass index (BMI), and evaluate the barriers encountered and the effect on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and understand English
* BMI ≥ to 25.

Exclusion Criteria:

* Regularly skip meals.
* Are unwilling or unable to limit eating to an 8-hour window.
* Have a current Melanoma or cancer diagnosis.
* Currently breastfeeding.
* Pregnant, or planned to be pregnant within 3 months.
* Are taking insulin or sulfonylurea drugs.
* Are taking weight loss medications or had weight loss surgery within the last year.
* Have a history of eating disorders.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in weight | Baseline, 12 weeks
  Reported in kilograms (kg)

SECONDARY OUTCOMES:
Change in Hemoglobin A1c | Baseline, 12 weeks
  Hemoglobin is a protein within red blood cells. As glucose enters the bloodstream, it binds to hemoglobin, or glycates. The more glucose that enters the bloodstream, the higher the amount of glycated hemoglobin. An A1C level below 5.7 percent is considered normal. Reported as percentage of glycated hemoglobin
Change in fasting glucose | Baseline, 12 weeks
  Glucose (sugar) measured in the blood and reported in milligrams per deciliter (mg/dL).
Change in total cholesterol | Baseline, 12 weeks
  Blood sample taken to measure the sum of blood's cholesterol content and reported in milligrams/deciliter (mg/dL)
Change in Low-density lipoprotein (LDL) cholesterol | Baseline, 12 weeks
  LDL (bad) cholesterol measured in the blood and reported in milligrams/deciliter (mg/dL)
Change in High-density lipoprotein (HDL) cholesterol | Baseline, 12 weeks
  HDL (good) cholesterol measured in the blood and reported in milligrams/deciliter (mg/dL)
Change in Triglycerides | Baseline, 12 weeks
  Triglycerides levels measured in the blood and reported in milligrams/deciliter (mg/dL)
Subjects to complete study | Baseline, 12 weeks
  Total number of subjects to complete study per protocol

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Bohn, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials